CLINICAL TRIAL: NCT04101916
Title: Paired Associative Stimulation in Subacute Spinal Cord Injury
Brief Title: PAS in Subacute SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anastasia Shulga, Principle Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WFL-FI-15/19
Record Dates: First submitted 2019-09-18; First posted 2019-09-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Intervention Model Description: The aim is 20 participants and the anticipated dropout percentage is 20%, therefore maximum number of randomized patients will be 24. If there will be no dropouts, only 20 patients will be recruited.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paired Associative Stimulation (Experimental)
  Interventions: Device: Paired associative stimulation
- Sham (Sham Comparator)
  Interventions: Device: Sham paired associative stimulation

INTERVENTIONS:
Device: Paired associative stimulation — Paired associative stimulation (PAS) administered several times per week for 12 weeks to upper limbs. PAS comprises transcranial magnetic stimulation (eXimia magnetic stimulator, Nexstim Ltd, Helsinki, Finland) and peripheral nerve stimulation (given with Dantec Keypoint® electroneuromyography device (Natus Medical Incorporated, Pleasanton, CA, USA)).
  Arms: Paired Associative Stimulation
Device: Sham paired associative stimulation — Sham transcranial magnetic stimulation and sham peripheral nerve stimulation.
  Arms: Sham

SUMMARY:
The investigators have recently shown in incomplete SCI patients that long-term paired associative stimulation is capable of restoring voluntary control over some paralyzed muscles and enhancing motor output in the weak muscles. In this study, the investigators will administer long-term paired associative stimulation to patients with incomplete cervical level SCI at the subacute stage, and investigate its effectiveness for upper extremity rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. SCI caused by an external trauma or SCI caused by nontraumatic non-progressive disease of the spinal cord
2. Cervical level injury, tetraplegia
3. Time from injury/onset of symptoms 1-4 months
4. Medical condition stable
5. Residual neural connectivity in upper extremity: some voluntary activity in finger muscles or MEPs obtainable from distal hand muscles

Exclusion Criteria:

1. Diagnosed brain damage, visible in MRI or CT.
2. No activity in hands/fingers and no MEPs recorded from distal hand muscles.
3. Epilepsy
4. Metal inclusion in the head area
5. High intracranial pressure
6. Pacemaker
7. Implanted hearing device
8. Progressive diseases of spinal cord or brain (e.g. malignant tumors, degenerative diseases).
9. History of malignant tumor within the past 5 years.
10. Previous head or spinal cord injury affecting the motor performance of upper extremities.
11. Congenital anomaly in the anatomical structure of spinal canal/cord or dura.
12. Significant systemic disease or other condition that could cause neurological deficit, or may affect subject's capability to undergo investigation-related procedures.
13. Acute severe infection.
14. Contraindications for MRI.
15. Current severe psychiatric diseases.
16. Current chronic drug and/or alcohol abuse.
17. Pregnancy.
18. Severe emergency care polyneuropathy
19. Pressure ulcer affecting the subject's capability to undergo the procedure safely

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Daniels and Worthingham's Muscle Testing | Change from baseline score immediately after, 6 months after and 1 year after last stimulation session
  hand muscle strength is evaluated on 0-5 scale (0=no movement, 5=normal)
Spinal Cord Independence Measure (SCIM) | Change from baseline score immediately after, 6 months after and 1 year after last stimulation session
  standard SCIM evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- BioMag laboratory, Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Background] Tolmacheva A, Savolainen S, Kirveskari E, Lioumis P, Kuusela L, Brandstack N, Ylinen A, Makela JP, Shulga A. Long-Term Paired Associative Stimulation Enhances Motor Output of the Tetraplegic Hand. J Neurotrauma. 2017 Sep 15;34(18):2668-2674. doi: 10.1089/neu.2017.4996. Epub 2017 Jul 21. PMID 28635523
- [Background] Shulga A, Lioumis P, Zubareva A, Brandstack N, Kuusela L, Kirveskari E, Savolainen S, Ylinen A, Makela JP. Long-term paired associative stimulation can restore voluntary control over paralyzed muscles in incomplete chronic spinal cord injury patients. Spinal Cord Ser Cases. 2016 Jul 14;2:16016. doi: 10.1038/scsandc.2016.16. eCollection 2016. PMID 28053760
- [Background] Tolmacheva A, Makela JP, Shulga A. Increasing the frequency of peripheral component in paired associative stimulation strengthens its efficacy. Sci Rep. 2019 Mar 7;9(1):3849. doi: 10.1038/s41598-019-40474-0. PMID 30846765
- [Background] Shulga A, Lioumis P, Kirveskari E, Savolainen S, Makela JP, Ylinen A. The use of F-response in defining interstimulus intervals appropriate for LTP-like plasticity induction in lower limb spinal paired associative stimulation. J Neurosci Methods. 2015 Mar 15;242:112-7. doi: 10.1016/j.jneumeth.2015.01.012. Epub 2015 Jan 15. PMID 25597909
- [Background] Shulga A, Zubareva A, Lioumis P, Makela JP. Paired Associative Stimulation with High-Frequency Peripheral Component Leads to Enhancement of Corticospinal Transmission at Wide Range of Interstimulus Intervals. Front Hum Neurosci. 2016 Sep 23;10:470. doi: 10.3389/fnhum.2016.00470. eCollection 2016. PMID 27721747
- [Background] Tolmacheva A, Savolainen S, Kirveskari E, Brandstack N, Makela JP, Shulga A. Paired associative stimulation improves hand function after non-traumatic spinal cord injury: A case series. Clin Neurophysiol Pract. 2019 Aug 13;4:178-183. doi: 10.1016/j.cnp.2019.07.002. eCollection 2019. PMID 31886442
- [Background] Rodionov A, Savolainen S, Kirveskari E, Makela JP, Shulga A. Restoration of hand function with long-term paired associative stimulation after chronic incomplete tetraplegia: a case study. Spinal Cord Ser Cases. 2019 Oct 1;5:81. doi: 10.1038/s41394-019-0225-5. eCollection 2019. PMID 31632739